CLINICAL TRIAL: NCT00663091
Title: A Prospective, Randomized Double-Blind Controlled Study of WPP-201 for the Safety and Efficacy of Treatment of Venous Leg Ulcers
Brief Title: A Prospective, Randomized, Double-Blind Controlled Study of WPP-201 for the Safety and Efficacy of Treatment of Venous Leg Ulcers
Acronym: WPP-201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 56-RW-001
Record Dates: First submitted 2008-04-18; First posted 2008-04-22 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Venous Leg Ulcers
Keywords: WPP-201

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bacteriophages (Experimental)
  Interventions: Drug: Bacteriophage; Drug: WPP-201 Bacteriophage; Drug: Bacteriophages

INTERVENTIONS:
Drug: Bacteriophage — WPP-201 is a pH neutral, polyvalent phage preparation, which contains 8 bacteriophages ("component bacteriophages" or "component phages") lytic for P. aeruginosa, S. aureus, and E. coli (Table 1). The cocktail contains a concentration of approximately 1 x 109 PFU/ml of each of the component monophages. The phage component of WPP-201 is roughly estimated to be £ 0.5 ppm by weight and the remainder is phosphate-buffered saline containing < 1,000 ppm total organic carbon from the growth medium and biomass. All phages contained in the preparation have been originally isolated from the environment, and they have not been genetically manipulated in any way (i.e., the preparation is 100% natural). WPP-201 contains no preservatives and antioxidants.
  Other Names: WPP-201- Bacteriophage
Drug: WPP-201 Bacteriophage — WPP-201 is a pH neutral, polyvalent phage preparation, which contains 8 bacteriophages ("component bacteriophages" or "component phages") lytic for P. aeruginosa, S. aureus, and E. coli (Table 1). The cocktail contains a concentration of approximately 1 x 109 PFU/ml of each of the component monophages. The phage component of WPP-201 is roughly estimated to be £ 0.5 ppm by weight and the remainder is phosphate-buffered saline containing < 1,000 ppm total organic carbon from the growth medium and biomass. All phages contained in the preparation have been originally isolated from the environment, and they have not been genetically manipulated in any way (i.e., the preparation is 100% natural). WPP-201 contains no preservatives and antioxidants.
  Other Names: WPP-201
Drug: Bacteriophages — WPP-201 is a pH neutral, polyvalent phage preparation, which contains 8 bacteriophages ("component bacteriophages" or "component phages") lytic for P. aeruginosa, S. aureus, and E. coli (Table 1). The cocktail contains a concentration of approximately 1 x 109 PFU/ml of each of the component monophages. The phage component of WPP-201 is roughly estimated to be £ 0.5 ppm by weight and the remainder is phosphate-buffered saline containing < 1,000 ppm total organic carbon from the growth medium and biomass. All phages contained in the preparation have been originally isolated from the environment, and they have not been genetically manipulated in any way (i.e., the preparation is 100% natural). WPP-201 contains no preservatives and antioxidants.

SUMMARY:
To test safety and efficacy of Bacteriophage on Venous Leg Ulcers.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled double blind study in patients with full thickness venous leg ulcers of greater than 30 days duration evaluating the safety of WPP-201 on the healing of those wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have evidence of hemosiderosis, stasis dermatitis, or dermato liposclerosis; AND edema in the lower extremity on which the wound is present.
2. Subject must be at least 18 years of age.
3. Subject must have a minimum life expectancy of at least 1 year to be determined by the Investigator.
4. The post-debridement ulcer at Day 0 must be free of all necrotic tissue and undermining.
5. The study ulcer must be from 1 cm2 to 60 cm2 in size.
6. The study ulcer must have been present for greater than 30 days at study Day -7.
7. The study ulcer is separated at least 4 cm from all other ulcers at Study Day -7 and Study Day 0 and has a margin of intact skin sufficient for anchoring of the required study dressings.
8. The subjects' Glycosylated hemoglobin (HbA1C) must be equal to or less than 10.0% for subjects with diagnosed diabetes at study Day 0.
9. The subject, legal guardian or authorized representative must have understood, signed and dated the IRB approved informed consent form.
10. The subject must be available for evaluation on a weekly basis for the twelve (12) weeks of the study. Visits at Week 13 and Week 14 are required for initial wound healing, which is achieved in study Week 11 or 12. The Investigator will evaluate both groups at Week 16 and Month 6. Subjects must be available for evaluation at Week 16 and Month 6.
11. Subjects' TCpO2 must be equal to or greater than 20 mm of mercury and ABI greater than 0.7.

Exclusion Criteria:

1. Subject whose ulcer has healed 30% or greater from the evaluation Study day -7 to the post-debridement Study Day 0 as determined by wound tracings using VisitrakTM.
2. A history of alcohol or substance abuse, within the previous year, which could, or in the judgment of the Investigator, would interfere with study compliance or protocol requirements.
3. Participation in clinical trials evaluating investigational pharmaceuticals or biologics within 3 months or devices within 30 days of admission to the study.
4. Subject with a history of receiving any of the following within the last 30 days: systemic corticosteroids exceeding a total daily dose of 20mg, immunosuppressive agents, radiation therapy or chemotherapy. Anticipated use of the above during the study period will also exclude a subject from entry into the study. Topical and inhaled corticosteroids are not prohibited.
5. Subject will be excluded if:

   * Serum sodium is less than 130 or greater than 147
   * Potassium is greater than 5.4 or less than 3.3
   * Glucose is less than 55
   * Blood urea nitrogen is greater than 31
   * Creatinine is greater than 2.1
   * Calcium is less than 7
   * CPK is greater than 3 times upper limits of normal
   * Albumin is less than 2.5
   * Total protein is less than 5
   * Alkaline phosphatase is greater than 3 times upper limits of normal
   * ALT/AST is greater than 5 times upper limits of normal
   * Hemoglobin is less than 8
   * White blood count is greater than 20,000 or below 1,000
6. Subject who is pregnant, lactating or has a positive serum hCG as determined by laboratory testing is excluded from the study.
7. Subject who demonstrates allergies to any component in WPP-201 (phage or saline).
8. Subject who has previously received any application of bacteriophage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2006-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of this Phase 1 study is to evaluate the safety of the use of WPP-201. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southweast Regional Wound Care Center, Lubbock, Texas, United States